CLINICAL TRIAL: NCT03526653
Title: Physical and Cognitive Exercises in Nursing Homes: Is Frailty Reversible?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Dominique Hansen, Principal Investigator, Hasselt University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: PAIE-001
Record Dates: First submitted 2018-04-21; First posted 2018-05-16 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Physical Activity; Elderly
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention 1 (Other): exercise on an ergometer or motomed in an environment without other visual stimuli
  Interventions: Other: exercise without visual stimuli
- Intervention 2 (Other): exercise on an ergometer or motomed while watching the National Geografics channel on television
  Interventions: Other: excercise with National Geografics
- Intervention 3 (Other): exercise on an ergometer or motomed with the interactive software program MemoRide with which participants can exercise in real life on a virtual manner
  Interventions: Other: Exercise with MemoRide
- Control group (No Intervention): Rest during 30 minutes

INTERVENTIONS:
Other: exercise without visual stimuli — exercise on an ergometer or motomed in an environment without other visual stimuli
  Arms: Intervention 1
Other: excercise with National Geografics — exercise on an ergometer or motomed while watching the National Geografics channel on television
  Arms: Intervention 2
Other: Exercise with MemoRide — excercise on an ergometer or motomed with the interactive software program MemoRide with which participants can exercise in real life on a virtual manner
  Arms: Intervention 3

SUMMARY:
Elderly in residential care spend 97% of their time sedentary. Moreover, exercise therapy often takes place in a poorly stimulating environment which is less motivational for the elderly to undertake regularly. Exercise is however necessary to preserve their physical capabilities and to limit their care dependence.

The aim of this study is to investigate the most motivating and stimulating exercise modality for prefrail and frail elderly in nursing homes with which they can reach sufficient training volume.

To study this, elderly will exercise in 3 different ways on an ergometer or motomed (according to their physical capabilities): 1) in an environment without other visual stimuli 2) in front of a television with National Geographic images 3) with the interactive software program MemoRide with which participants can exercise in real life on a virtual manner.

MemoRide (Activ84Health) uses Google Street View images. The starting point is a connection between an exercise bike and a tablet with a pedalling sensor. This way, pedal frequency is sent to the tablet and as a result, images continue when pedalling.

The forth modality is the control modality, in which participants are instructed to rest (supine) during 30 minutes.

Based on objective training parameters and metabolic parameters e.g. glucose, insulin, brain-derived neurotrophic factor (BDNF) and lactate, (via a blood sample with a venous catheter) the training modality which offers the best training results will be studied. Secondly, also subject experiences (motivation and emotions) will be evaluated by using questionnaires and observation scales.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with an age of at least 70 years at the start of the study;
* Staying for at least one month in WZC St. Elisabeth Hasselt at the start of the study;
* Being frail or prefrail (according to the criteria of Fried);
* Being available to participate in the study during 4 consecutive weeks;
* Being able to actively exercise on an exercise bike (if necessary from a wheelchair) during at least 5 minutes;
* Understand simple instructions.

Exclusion Criteria:

* Any neurological or orthopedic disease which makes it impossible to exercise by bike actively e.g. stroke with hemiparesis of the lower limbs, amputations of the lower limbs,…;
* Any disease which makes it impossible to exercise actively e.g. heart failure;
* Any neurological or orthopedic disease from which progression (e.g. hip prosthesis, acute stroke) due to active recovery or decline (e.g. ALS (amyotropic lateral sclerosis), MS) due to the disease process can be expected on short term (1-2 months);
* Being blind or visually impaired;
* Any acute disease on the moment of the intervention which makes it impossible to exercise by bike during 30 minutes (e.g. hyper- or hypoglycemia) (reported by the caregiver)

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Brain Derived Neurotrophic Factor (BDNF) | Baseline
  a protein produced inside the brain which can be transported outside the brain - it probably has a protective effect on neuronal survival and maintenance during adulthood
Brain Derived Neurotrophic Factor (BDNF) | minute 30
  a protein produced inside the brain which can be transported outside the brain - it probably has a protective effect on neuronal survival and maintenance during adulthood
Distance immediately post-intervention | minute 30
  evaluation of distance via data on the exercise bike
Velocity | minute 30
  evaluation of velocity via data on the exercise bike and pedalling sensor
Intrinsic Motivation Inventory | minute 30
  evaluation of motivation via Intrinsic Motivation Inventory questionaire
Observed Emotion Rating Scale | minute 30
  evaluation of emotions via an observation scale (Observed Emotion Rating Scale)
Fatigue | minute 30
  evaluation of perceived exertion via the BORG-scale
Credibility-Expectancy Questionnaire | minute 30
  evaluation of motivation via Credibility-Expectancy Questionnaire

SECONDARY OUTCOMES:
Glucose | baseline
  Evaluation of glucose via a blood sample
Glucose | minute 30
  Evaluation of glucose via a blood sample
Insulin | baseline
  Evaluation of insulin via a blood sample
Insulin | minute 30
  Evaluation of insulin via a blood sample
Heart rate | baseline
  Evaluation of heart rate via a heart rate monitor
Heart rate | minute 30
  Evaluation of heart rate via a heart rate monitor
systolic and diastolic blood pressure | baseline
  Evaluation of blood pressure via a blood pressure monitor
systolic and diastolic blood pressure | minute 30
  Evaluation of blood pressure via a blood pressure monitor
Lactate | minute 30
  Evaluation of lactate via a finger prick
depressed feelings | baseline
  Evaluation of depressed feelings via a questionnaire (Geriatric Depression Scale)

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Hansen, prof. dr., Principal Investigator — Hasselt University; Nastasia Marinus, drs., Study Chair — Hasselt University
Locations (1):
- WZC Begralim (Campus Sint-Elisabeth), Hasselt, Belgium